CLINICAL TRIAL: NCT03676738
Title: Cohort Study of Risk Factors for Postoperative Cognitive Decline
Acronym: POCD
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Katie J. Schenning, Principal Investigator, Oregon Health and Science University
Other Study IDs: 17595
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Decline
Keywords: Anesthesia, Risk Factors, Age
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained for DNA extraction and storage. Genotyping will be done in batches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In-patient spine surgery: Scheduled for an in-patient, elective spine surgery where subject will receive general anesthesia
- Non-surgical spine care: Presenting to spine clinic and undergoing conservative, non-surgical management of spine disorder

SUMMARY:
Presently, the role of either genetic factors or biological sex in the development of postoperative cognitive dysfunction (POCD) is unknown. There is a critical need to determine which individuals are at high-risk for developing POCD by virtue of biological sex or genetic predisposition. The knowledge gained in the described research has the potential to shed light on mechanistic pathways, a necessary next step in order to ultimately identify therapeutic strategies.

DETAILED DESCRIPTION:
Adults 65 years and older represent the fastest-growing age group in the United States, and account for one third of all surgical patients. These older adults are at the highest risk for deleterious postoperative neurocognitive outcomes. Postoperative cognitive dysfunction (POCD) occurs in up to 40% of older adults after major non-cardiac surgery. POCD is a syndrome characterized by a decrease in performance on neuropsychological test battery from before to after surgery. Neuropsychological testing for POCD typically spans cognitive domains including memory, attention, concentration, and/or executive function. There is an increasing body of literature suggesting that exposure to surgery and anesthesia increases the risk of Alzheimer's disease (AD). Surgery and anesthesia enhance neuropathologic changes known to underlie AD including amyloid beta accumulation and aggregation, neuroinflammation, increased levels of tau and tau phosphorylation, and memory decline. However, not everyone with a history of surgery and anesthesia develops POCD, suggesting biological risk factors are involved.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an in-patient, elective spine surgery where subject will receive general anesthesia
* Presenting to spine clinic and undergoing conservative, non-surgical management of spine disorder
* Subjects must have sufficient vision and hearing to complete neuropsychological testing
* Proficient in spoken and written English language

Exclusion Criteria:

* Diagnosed dementia or dementia-related treatment (i.e. donepezil prescription, or memory-care facility residence)
* Significant disease of the central nervous system (CNS) (i.e. Parkinson's disease)
* History of stroke or traumatic brain injury
* Major psychiatric disorder (i.e. schizophrenia)
* Alcohol or drug abuse according to DSM-V within the last 2 years
* Need for urgent/emergent surgery
* Surgery/anesthesia within prior 12 months
* Refusal of consent

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects who present to spine clinic
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Genetic Variables | Six months
  To determine whether specific genetic variables (i.e. APOE4 or PLA2 alleles) and/or biological sex confer a higher risk to developing postoperative cognitive and functional status decline in older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Schenning, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States